CLINICAL TRIAL: NCT06349902
Title: Re-linking People With Diagnosed But Untreated HCV to Care in a Community-based Substance-use Telemedicine Program
Brief Title: Re-link HCV in Substance-Use Telemedicine Program
Status: Recruiting | Type: Observational
Sponsor: trueNorth Medical Centres (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00077561
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Positive HCV RNA, no sufficient previous course of DAA treatment.: Having a positive HCV RNA laboratory result and lacking a sufficient previous course of DAA treatment.
  Interventions: Behavioral: Re-Link

INTERVENTIONS:
Behavioral: Re-Link — The HCV nurse will attempt to contact the PWDU HCV via phone call and text. If unable to connect with a client via phone, an alert is added to the client's chart in the electronic medical record. When the client presents to the CBSUTP for their regular substance use follow up appointment, the chart alert is flagged by the administrative team and the client is connected with the HCV nurse via telemedicine. Clients who are connected to the HCV team are considered re-linked. The HCV nurse will provide an HCV intake as per program guidelines. Clients who would prefer to pursue treatment elsewhere will be supported with a referral to their family doctor or an alternative HCV program in the community. Clients who choose to be treated at the CBSUTP will receive a HCV consultation, DAA treatment and follow-up from the HCV clinical team onsite as per existing program guidelines.

SUMMARY:
This is an observational, retrospective & prospective cohort study. The retrospective element of the study is a chart review to identify people with diagnosed but untreated HCV and re-link them to care. The observational prospective cohort element of the study will examine the HCV linkage to care, treatment initiation, treatment completion & cure rates of these HCV clients achieved through this chart review and re-linking approach.

DETAILED DESCRIPTION:
The study, led by trueNorth medical center in Ontario, focuses on re-linking people diagnosed with untreated Hepatitis C (HCV) to care through a community-based substance-use telemedicine program. HCV is a significant health concern in Canada, especially among people who inject drugs (PWID), who face barriers to accessing treatment. Integrating HCV treatment with substance use care may improve treatment uptake.

This observational study includes both retrospective and prospective cohorts. The retrospective aspect involves chart reviews to identify untreated HCV patients for re-linking, while the prospective cohort examines treatment outcomes such as linkage to care and cure rates. Participants include individuals over 18 with a positive HCV RNA result who have not completed a course of Direct-Acting Antiviral (DAA) treatment. Excluded are those unable to consent or with restricted access to their health records.

Study procedures involve identifying untreated HCV patients, attempting re-linkage via telecommunication, and offering treatment through the program. Outcome measures include the number of patients re-linked to care and their treatment outcomes. Data analysis will utilize IBM SPSS for logistic regression and descriptive statistics, aiming to evaluate the efficacy of this telemedicine approach in improving HCV care among PWID.

Ethical considerations include informed consent and data privacy, with oversight by the ADVARRA Canadian Institutional Review Board. The study seeks to address HCV care gaps in PWID populations by leveraging telemedicine for improved access and treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

For the retrospective chart review element of the study, inclusion criteria includes anyone who had a telemedicine visit at the community based substance use telemedicine program between January 1st 2023 and December 31st 2024.

For the prospective cohort element of the study, the inclusion criteria are listed below:

Aged ≥18. Ability and willingness of the participant to provide informed consent. Having a positive HCV RNA laboratory result and lacking a sufficient previous course of DAA treatment.

Exclusion Criteria:

For the retrospective chart review element of the study, exclusion criteria is: a consent directive to restrict access to their OLIS record.

For the prospective cohort study, exclusion criteria is an inability or unwillingness of the participant to provide informed consent.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population for this research comprises individuals diagnosed with Hepatitis C Virus (HCV) who have not yet received treatment. Key characteristics of the study population include:
  Age: Participants are aged 18 years or older. Health Condition: All individuals have a confirmed positive HCV RNA laboratory result, indicating an active HCV infection but lack a sufficient previous course of treatment with Direct-Acting Antivirals (DAAs).
  Telemedicine Engagement: They have had at least one telemedicine visit with the community-based substance use telemedicine program (CBSUTP) between January 1st, 2023, and December 31st, 2024.
  Informed Consent: Participants possess the ability and willingness to provide informed consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
number of patients identified as having diagnosed but untreated HCV | March 2024 - August 2024
  number of patients identified as having diagnosed but untreated HCV
percentage of patients identified as having diagnosed but untreated HCV that are re-linked to HCV care | March 2024 - December 2024
  percentage of patients identified as having diagnosed but untreated HCV that are re-linked to HCV care

SECONDARY OUTCOMES:
treatment initiation rates | March 2024 - December 2024
  treatment initiation rates
treatment completion dates | March 2024 - December 2024
  treatment completion dates
cure rates | March 2024 - December 2024
  cure rates

CONTACTS AND LOCATIONS:
Overall Officials: Hannah O'Reilly, Study Director — trueNorth Medical
Locations (1):
- trueNorth Medical Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No